CLINICAL TRIAL: NCT00871663
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of the Cyclin-Dependent Kinase (CDK) Inhibitor SCH 727965 Administered Weekly in Subjects With Advanced Malignancies
Brief Title: Phase 1 Weekly Dosing of SCH 727965 in Patients With Advanced Cancer (Study P04629AM6)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04629
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Solid Tumors; Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Lymphocytic, Chronic. B-Cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, B-Cell | interventions — dinaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Advanced solid tumors (Experimental): Participants with advanced solid tumors treated with SCH 727965 in dose-escalation cohorts
  Interventions: Drug: SCH 727965
- Non-Hodgkin's lymphoma and multiple myeloma (Experimental): Participants with non-Hodgkin's lymphoma or multiple myeloma treated with SCH 727965
  Interventions: Drug: SCH 727965
- B cell chronic lymphocytic leukemia (Experimental): Participants with B-cell chronic lymphocytic leukemia treated with SCH 727965 in dose-escalation cohorts
  Interventions: Drug: SCH 727965

INTERVENTIONS:
Drug: SCH 727965 — Dose escalation of SCH 727965 IV administered in 28-day cycles, on Days 1, 8, and 15 of each 28-day cycle.

SUMMARY:
The study will evaluate the safety, tolerability, maximum administered dose, and dose limiting toxicity of SCH 727965 administered as an intravenous infusion on Days 1, 8 and 15 of each 28 day cycle in participants with solid tumors, non Hodgkins lymphoma, multiple myeloma or chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years, either sex, any race.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
* There must be no known standard therapy, or disease must be refractory to standard therapy
* Adequate hematologic, renal, and hepatic organ function and laboratory parameters
* For advanced solid tumors, non-Hodgkin's lymphoma, or multiple myeloma:

  * Participants must have histologically proven solid tumors, non-Hodgkin's lymphoma, or multiple myeloma.
  * Evaluable malignancy must be present by computed tomography or magnetic resonance imaging, obtained within 4 weeks prior to the start of treatment with SCH 727965.
* Subjects with multiple myeloma must have measurable disease defined as:

  * Serum monoclonal protein greater than 0.5 g/dL or urine light chain excretion of greater than 0.2 g/24-hour obtained within 4 weeks prior to the start of treatment.
  * Participants with lower M protein values or nonsecretory myeloma are eligible if measurable disease can be established within 4 weeks prior to start of treatment, such as:

    * serum free light chain ratio greater than 5 times the normal ratio limit; and/or
    * measurable soft tissue plasmacytoma greater than 2 cm, by either physical examination and/or applicable radiographs; and/or
    * bone marrow involvement greater than 30%.
* For B-cell chronic lymphocytic leukemia (B-CLL):

  * Diagnosis of B-CLL according to the National Cancer Institute Working Group (NCI-WG) criteria or a histological diagnosis of small lymphocytic lymphoma.
  * Disease must be evaluable according to NCI-WG response criteria.

Exclusion Criteria:

* Symptomatic brain metastases or primary central nervous system malignancy.
* Previous radiation therapy to >25% of the total bone marrow.
* Previous treatment with SCH 727965.
* Known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SCH 727965, including maximum administered dose and dose-limiting toxicity. | End of trial
In participants with advanced solid tumors, non Hodgkin's lymphoma or multiple myeloma, pharmacodynamic effects of SCH 727965 with an ex vivo lymphocyte stimulation assay of participant's peripheral blood lymphocytes. | End of trial

REFERENCES:
- [Background] Flynn J, Jones J, Johnson AJ, Andritsos L, Maddocks K, Jaglowski S, Hessler J, Grever MR, Im E, Zhou H, Zhu Y, Zhang D, Small K, Bannerji R, Byrd JC. Dinaciclib is a novel cyclin-dependent kinase inhibitor with significant clinical activity in relapsed and refractory chronic lymphocytic leukemia. Leukemia. 2015 Jul;29(7):1524-9. doi: 10.1038/leu.2015.31. Epub 2015 Feb 24. PMID 25708835
- [Result] Nemunaitis JJ, Small KA, Kirschmeier P, Zhang D, Zhu Y, Jou YM, Statkevich P, Yao SL, Bannerji R. A first-in-human, phase 1, dose-escalation study of dinaciclib, a novel cyclin-dependent kinase inhibitor, administered weekly in subjects with advanced malignancies. J Transl Med. 2013 Oct 16;11:259. doi: 10.1186/1479-5876-11-259. PMID 24131779